CLINICAL TRIAL: NCT05772936
Title: Perturbation-induced Reactive Standing BalanceTraining in Persons Post Stroke
Brief Title: Reactive Standing Balance Step Training Post Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Katherine Martinez, Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RST4CVA2018
Record Dates: First submitted 2019-10-24; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Stroke, Cerebrovascular
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm non-randomized (Experimental): all enrolled subjects will participate in the perturbation-induced step training, 1 or 6 sessions about 1-1.5 hour (30-90 trials) each session.
  Interventions: Behavioral: Balance training

INTERVENTIONS:
Behavioral: Balance training — perturbation induce step training to improve reactive stepping with paretic leg.

SUMMARY:
The purpose of this study is to investigate the effectiveness of reactive step training on the timing and frequency of perturbation induced paretic leg stepping in persons post stroke. The study will consist of one or six one-hour training sessions and a pre and post visit each lasting up to two hours at our downtown Chicago location.

DETAILED DESCRIPTION:
Perturbation induced step training. Perturbations will be applied by a mechanical weight drop system that has been used in previous studies. A belt with a cable will be attached to the subject's waist. The cable will be attached to metal weights that is held by an electromagnet on a vertical pole approximately 10-12ft from the subject. The weight will drop 52cm when the electromagnet is released. When the subject has attained and held a predetermined standing position for 1-3 seconds the mechanical perturbation will be activated. See training protocol below.

Pre and Post Testing Sessions: Subjects will be asked to complete pre and post testing sessions within 1 week of training. Testing sessions will include laboratory and clinical measures of balance and will last for approximately one hour.

Laboratory Measures: Participants will complete 2 standing trials, 12 voluntary stepping trials, and 12 anterior perturbation trials while standing on force platforms.

Standing trials: Subjects will be asked to stand feet hip with apart with each foot on a separate force plate that measure the pressure under their feet. Their foot placement will be traced so they can return to the same placement for each trial. Subjects will be instructed to cross their arms and stand as still as they can for 3 seconds, then march in place for 3 seconds.

Voluntary Stepping Trials: While standing with their feet in their foot tracings subjects will be asked to shift their weight until they assume a predetermined pressure under each foot. Visual feedback will be provided on a monitor in front of them. They will be instructed to hold that position until they see the "Go" cue on the screen at which point they should take 3 steps forward as fast as they can. There will be 6 stepping trials on each leg starting with the less involved leg.

Reactive Stepping Trials: Subjects will be secured in a safety harness that is mounted to the ceiling. The harness does not interfere with stepping but allows the person body weight to be supported if there is a loss of balance. A belt will be placed around the subjects' waist that will be connected by a cable to a mechanical weight drop device that will pull the subject forward to challenge their balance. The puller will provide mechanical perturbations up to 10% of subjects' body weight. The subjects will be instructed not resist the pull but to respond naturally and move their feet if needed to maintain up right posture. There will be ten reactive trials. Rest breaks will be given between voluntary and reactive trials or as needed.

Participants will complete 6 training sessions within a three-week period. Subjects will stand with their feet on a platform with a scale. Subjects will be instructed to try to use their more impaired leg if they need to step. The same mechanical perturbation that was used in the pre/post testing will be used for training with the belt attached to their waist. When they have attained and held a predetermined standing position for 1-3 seconds the mechanical perturbation will be activated. The weight bearing status of the more impaired leg will be increased by 5% after 10 out of 12 successive trials (i.e. stepping with the more impaired leg) or decreased by 5% if they always step with the less impaired leg after 6 trials. Training sessions will consist of 50 perturbation trials at 10% body weight and 3 catch trials at 2% body weight to discourage premature stepping. Training session will last about 1 hour. Subjects will be given rest breaks as needed.

ELIGIBILITY:
Inclusion Criteria:

1. at least 1 year post a single unilateral hemispheric stroke (CVA)
2. living independently in the community
3. able to walk 25 feet without assistive device

Exclusion Criteria:

1. pain that limits movement
2. joint surgery of the lower extremity
3. unable to give consent
4. significant postural alignment deficits such as scoliosis or genu recurvatum
5. loss of sensation in the lower limb

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Change in frequency of stepping with paretic leg after a perturbation | Change in stepping with paretic leg will be modeled from baseline and immediately after the intervention.
  number of trials when the paretic leg takes the first reactive step after the perturbation is applied during the reactive trials.
Change in step onset time for voluntary and reactive steps | Change in step onset will be modeled from baseline and immediately after the intervention.
  step onset time is the time the stepping foot lifts off the ground after the Go cue for voluntary steps and after the perturbation for the reactive steps.
Change in reactive lean balance test | Change in reactive lean balance test will be modeled from baseline and immediately after the intervention.
  Lean balance test is a passive way to test reactive stepping. Participants will lean again the research staff hands until their center of mass is at the edge of their feet. The research staff will suddenly remove their hands and allow the participant to catch their balance. Research staff are trained to perform the test and to guard the participant if needed. Extra personnel will be near by for additional support if the participant is not able to recover their balance.

SECONDARY OUTCOMES:
10 meter walk test | Day 1 before training
  subject walking will be timed at comfortable and fast speed over a 10 meter distance.
Activities-specific Balance Confidence scale (ABC) | Day 1 before training
  The ABC is a sixteen item questionnaire that ask subjects to rate their balance confidence on various daily activities. Scores range from 10 to 100 on each item, with total score the average of all responses. Higher score indicate more balance confidence, low score indicate less balance confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Martinez, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available 6 months after publication
Access Criteria: access to data will be made available by contacting the principle investigator.